CLINICAL TRIAL: NCT01314846
Title: Co-culture Versus Sequential Culture System in Advanced Maternal Age.
Brief Title: Co-culture and Advanced Maternal Age in PGS Program
Acronym: CC-PGS
Status: Terminated | Type: Observational
Why Stopped: difficulty to include patients
Sponsor: IVI Madrid (Other)
Responsible Party: Principal Investigator, Fernando Bronet, PhD, IVI Madrid
Other Study IDs: MAD-MN-10-2011-03
Record Dates: First submitted 2011-03-10; First posted 2011-03-15 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2011-03

CONDITIONS: Age Factors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Control Group: sequential culture system
- Co-culture system

SUMMARY:
Fertilization and embryo development in vivo occurs in appropriate conditions in the mammalian reproductive tract. However in assisted reproductive technology (ART) embryos and oocytes are exposed to certain factors such as temperature, O2 pressure and pH fluctuations that may affect embryo development and viability in vitro. In Preimplantation Genetic Screening program (PGS) the investigators need to culture the embryos until day 5 so the requirement of culture techniques must be optimal to produce acceptable blastocyst rates. As it has been shown before, embryo culture conditions have the potential to impact biopsied embryos and hence PGS success rates.

Nowadays the coculture system with endometrial cells could be an alternative option to improve the blastocyst rates since some publications have indicated that endometrial cells may provide trace elements and growth factors that are not present in defined culture media and reproduce physiologic conditions. Although the role of coculture in vitro fertilization (IVF) has been controversial, a recent meta-analysis has established the potential benefits of coculture system.

The aim of this study was to compare embryologic and clinical outcomes in terms of blastocyst, implantation and pregnancy rates to evaluate endometrial epithelial cell (EEC) coculture versus sequential culture system in advanced maternal age ( ≥39 years) in the PGS program.

ELIGIBILITY:
Inclusion Criteria:

* Advanced maternal age (>39) undergoing PGS cycle

Exclusion Criteria:

* Other PGS indication
* Altered karyotype

Ages: 40 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women over 39 years old undergoing a PGS cycle
Sampling Method: Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
implantation rate | from February 2009 to December 2010

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Madrid, Madrid, Madrid, Spain